CLINICAL TRIAL: NCT02094508
Title: Impact of Trimethoprim-sulfamethoxazole Prophylaxis on Malaria Infection and Immunity in Children in Uganda
Brief Title: Impact of TMP-SMX Prophylaxis on Malaria Infection and Immunity in Children in Uganda
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999914073; 14-I-N073
Record Dates: First submitted 2014-03-20; First posted 2014-03-21 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2016-12-14

CONDITIONS: Malaria
Keywords: Parasitemia; HIV-Exposed; HIV-Unexposed; Liver Stage; Randomized
MeSH Terms: conditions — Malaria; Parasitemia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

SUMMARY:
Background:

- Malaria is a disease that affects many children and adults in Uganda and Africa. If it is not treated, it can make some people severely ill. TMP-SMX (Trade names Bactrim, Septrin) is a drug that is given to children born to HIV-positive mothers to help prevent infection. Studies have shown that TMP-SMX also may kill malaria infection in the very early stages of infection in the body, which may positively impact the way the body can fight malaria infection. Researchers want to know if giving TMP-SMX for 6 months longer than usual helps children fight malaria better in this way.

Objective:

- To find out if taking TMP-SMX for longer than usual helps fight off malaria in infants.

Eligibility:

- Infants 0-6 weeks of age who are HIV negative.

Design:

* Infants will be screened with a medical history and physical exam. A small amount of blood will be taken. The mothers medical records will be reviewed. Mothers will be asked about when they breastfeed.
* Participants will take TMP-SMX according to their doctor s orders. In Uganda, mothers will get a mosquito net with insecticide on it as per standard of care.
* Participants will come to the clinic once a month, every month, until the study ends in 2 3 years. Each visit will repeat the screening visit.
* Participants will also visit the clinic every month for a medical history, physical exam, and different blood tests.
* Six weeks after breastfeeding is stopped, children taking TMP-SMX will come into the clinic and will either be taken off the drug or will continue taking the drug for 6 more months.
* If a child becomes sick, it is important that the mother bring him or her to the RHSP clinic in Rakai.

DETAILED DESCRIPTION:
Malaria remains one of the most significant causes of morbidity and mortality throughout the world. Recent studies indicate that drugs used in HIV management can have antimalarial properties. In animal models, prophylactic doses of trimethoprim-sulfamethoxazole (TMPSMX), an antibiotic commonly used as prophylaxis against opportunistic infections in HIVexposed and HIV-infected patients, have been shown to arrest liver stage development of malaria parasites. Indeed, the liver stage of malaria parasites may be important to target since it is during this stage that clinical symptoms are absent and fewer parasites are present. TMP-SMX, used in HIV-exposed and HIV-infected subjects for opportunistic infection prophylaxis, significantly reduces clinical malaria, even in areas of moderate to high transmission intensity and high antifolate drug resistance. It is possible that reduction in liver stage parasite burden contributes to this unexpected effect. Nonetheless, the contribution of this liver-stage parasite killing to the reduction in clinical malaria observed in patients receiving TMP-SMX remains undescribed. Our primary objective aims to answer whether TMP-SMX reduces liver stage malaria infection.

For our exploratory objectives, we are interested in TMP-SMX effects on the development of anti-infection malaria immunity and effects on transmission. In mice, TMP-SMX prophylaxis during repeated malaria exposures has been shown to induce protective, anti-infection immunity against malaria (Charlotte Hobbs, unpublished data), which is distinct from naturally acquired immunity in which, after multiple infections, patients have less severe disease. TMP-SMX impact on the development of malaria-specific immunity, however, requires further investigation. Also, TMP-SMX has been shown to have sporonticidal (mosquito-oocyst killing) activity at levels achieved in patients on TMP-SMX prophylaxis in susceptible strains of P. falciparum, but the effects of TMP-SMX on transmission in the field remain undescribed.

This randomized study plans to enroll 164-220 HIV-uninfected, HIV-exposed (HUE) and 60 HIV-uninfected, HIV-unexposed (HUU) children in Kalisizo Hospital Health Center, Labor and Delivery Unit, Kalisizo, located within Rakai District, Uganda. HUE children will be randomized 1:1 into 2 arms. In the first arm (Standard of Care [SOC] arm), 82-110 children will receive TMP-SMX until 6 weeks after cessation of breast-feeding (age 12-18 months). In the second arm (Extended Prophylaxis [EP] arm), 82-110 children will receive SOC and remain on TMP-SMX for an additional 6 months after the cessation of breast-feeding. The 60 HUU children will serve as controls to establish baseline infection parameters in the community. Blood will be drawn from all subjects monthly via heel/finger stick to analyze malaria parasitemia. Additionally, venous blood will be drawn every 6 months to analyze cellular and humoral immunity. The duration of this study participation will be a minimum of 2 and up to 3 years.

Assessment of TMP-SMX impact on liver stage malaria infection and the development of protective anti-infection immunity in children will help guide decisions regarding TMP-SMX prophylaxis duration for HIV-exposed children in malaria endemic areas.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Infant must be born during the period beginning May 1, 2014 and ending November 30, 2014.
  2. Mothers of HUE subjects must be giving their child TMP-SMX prophylaxis at screening (this does not apply to HUU subjects).
  3. Mothers must be breastfeeding their child at screening.
  4. Parent/legal guardian must be able and willing to provide signed informed consent on behalf of the child subject, agree to bring the child to the study site for visits, and seek medical care for intercurrent illness for the child subject at the study site.
  5. Parent/legal guardian of HUE subjects must agree to be compliant with administering the daily prophylactic doses of TMP-SMX according to the standard guidelines.
  6. Mothers must consent to a review of their medical records and a monthly assessment of breastfeeding status.
  7. Mother/guardian must live within the Rakai District.

EXCLUSION CRITERIA:

1. Child has a diagnosis of HIV-infection or clinical or laboratory evidence of other chronic infection or disease (including renal or hepatic insufficiency).
2. Clinical determination of conditions that would exclude the child

   based on record review, history, and examination.
3. Participation in a malaria vaccine study or have a history of

involvement in such a study.

Ages: 2 Months to 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 173 (Actual)
Dates: Start 2014-03-07; Primary Completion 2015-12-28 (Actual); Study Completion 2016-12-14 (Actual)

PRIMARY OUTCOMES:
Malaria incidence rate (number of new malaria parasitemia episodes per time at risk) in HUE children on TMP-SMX prophylaxis compared to HUU children (not on TMP-SMX prophylaxis) between enrollment and study end. A malaria parasitemia episode is ... | At end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Steven J Reynolds, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- Rakai Health Sciences Program Uganda Virus Research Institute, Kalisizo, Uganda

REFERENCES:
- [Background] Mutanga JN, Raymond J, Towle MS, Mutembo S, Fubisha RC, Lule F, Muhe L. Institutionalizing provider-initiated HIV testing and counselling for children: an observational case study from Zambia. PLoS One. 2012;7(4):e29656. doi: 10.1371/journal.pone.0029656. Epub 2012 Apr 20. PMID 22536311
- [Background] Flateau C, Le Loup G, Pialoux G. Consequences of HIV infection on malaria and therapeutic implications: a systematic review. Lancet Infect Dis. 2011 Jul;11(7):541-56. doi: 10.1016/S1473-3099(11)70031-7. PMID 21700241
- [Background] Hobbs CV, Voza T, Coppi A, Kirmse B, Marsh K, Borkowsky W, Sinnis P. HIV protease inhibitors inhibit the development of preerythrocytic-stage plasmodium parasites. J Infect Dis. 2009 Jan 1;199(1):134-41. doi: 10.1086/594369. PMID 19032102
- [Derived] Kasule J, Gabriel EE, Anok A, Neal J, Eastman RT, Penzak S, Newell K, Serwadda D, Duffy PE, Reynolds SJ, Hobbs CV. Sulfamethoxazole Levels in HIV-Exposed Uninfected Ugandan Children. Am J Trop Med Hyg. 2018 Jun;98(6):1718-1721. doi: 10.4269/ajtmh.17-0933. Epub 2018 Apr 19. PMID 29692311